CLINICAL TRIAL: NCT01062243
Title: Brain Injury Inpatient Educational Intervention for Families and Caregivers (a Research Project Within the Traumatic Brain Injury Model System)
Brief Title: Brain Injury Inpatient Educational Intervention for Families and Caregivers
Acronym: BIIG-FACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H133A070036
Record Dates: First submitted 2010-01-29; First posted 2010-02-04 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Traumatic Brain Injury; Acquired Brain Injury
Keywords: brain injury; family treatment
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain Injury Education (Experimental): The Brain Injury Inpatient Guide for Families and Caregivers (BIIG-FACS), developed by J. Niemeier and J. Kreutzer, is a comprehensive intervention to meet the needs of family members and significant others of patients who are undergoing acute brain injury rehabilitation.
  Interventions: Behavioral: Brain Injury Education

INTERVENTIONS:
Behavioral: Brain Injury Education — The Brain Injury Inpatient Guide for Families and Caregivers (BIIG-FACS), developed by J. Niemeier and J. Kreutzer, is a comprehensive intervention to meet the needs of family members and significant others of patients who are undergoing acute brain injury rehabilitation.

SUMMARY:
The Brain Injury Inpatient Guide for Families and Caregivers (BIIG-FACS) is a comprehensive intervention to meet the needs of family members and significant others of patients who are undergoing acute, inpatient brain injury rehabilitation.

DETAILED DESCRIPTION:
The Brain Injury Inpatient Guide for Families and Caregivers (BIIG-FACS), developed by J. Niemeier and J. Kreutzer, is a comprehensive intervention to meet the needs of family members and significant others of patients who are undergoing acute brain injury rehabilitation. Program development was guided by considerable clinical experience, research review, and solicited consumer feedback.

The intervention has been manualized to facilitate efficient and effective administration. Now, a rigorous investigation involving randomized assignment to treatment and control groups is needed to empirically examine outcomes. Helping family members to cope more effectively has the potential to improve outcomes for persons with ABI. Strengthening families can enable persons with ABI to live more independently, achieve greater community integration, and live healthier lives. The investigation serves as a logical next step forward in advancing our understanding of standardized interventions designed to serve the family unit.

ELIGIBILITY:
Inclusion Criteria:

* Family members/caregiver friends of patients with ABI will be eligible to participate in the present investigation. ABI is defined as damage to brain tissue caused by stroke, aneurysm, anoxia, non-progressive brain tumor, infection, or an external mechanical force as evidenced by: loss of consciousness, post traumatic amnesia (PTA), objective neurological findings, or skull fracture.
* Lacerations and/or bruises of the scalp or forehead without other criteria listed above will be excluded.
* All family member participants and patients must be at least 18 years of age or older and able to understand and provide consent (or assent in the case of the patients).

Exclusion Criteria:

* Family members at imminent risk of psychiatric hospitalization, or in imminent danger of hurting themselves or others, as judged by the investigators, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Knowledge gained from educational materials | Post-treatment and 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Kreutzer, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Niemeier JP, Kreutzer JS, Marwitz JH, Sima AP. A Randomized Controlled Pilot Study of a Manualized Intervention for Caregivers of Patients With Traumatic Brain Injury in Inpatient Rehabilitation. Arch Phys Med Rehabil. 2019 Apr;100(4S):S65-S75. doi: 10.1016/j.apmr.2018.07.422. Epub 2018 Jul 31. PMID 30075147